CLINICAL TRIAL: NCT04089696
Title: Validation of the "Exspiron©" in Patients With Amyotrophic Lateral Sclerosis; Non-invasive Monitoring of Respiratory Volume.
Brief Title: Validation of the "ExSpiron©" in Patients With ALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Peter Wijkstra, Principal Investigator P.J. Wijkstra, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UMCG
Record Dates: First submitted 2019-09-06; First posted 2019-09-13 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Amyotrophic Lateral Sclerosis; Neuromuscular Diseases
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: Intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ExSpiron (Experimental): 10 patients with ALS
  Interventions: Device: ExSprion

INTERVENTIONS:
Device: ExSprion — The primary objective is the validation of the ExSpiron© non-invasive monitor in patients diagnosed with ALS.

SUMMARY:
Non-invasive ventilation (NIV) in patients diagnosed with amyotrophic lateral sclerosis (ALS) is nowadays common practice to provide comfort at the end stage of the disease. As complaints vary there is the need of a non-invasive device to measure respiratory volume to objectify complaints.

The ExSpiron© is a device for non-invasive monitoring of respiratory volume. The validation of this monitor in patients with ALS is the aim of this study.

The hypothesis is that the ExSpiron© delivers a valid assessment of respiratory volume in patients with ALS

DETAILED DESCRIPTION:
Rationale: Non-invasive ventilation (NIV) in patients diagnosed with amyotrophic lateral sclerosis (ALS) is nowadays common practice to provide comfort at the end stage of the disease. As complaints vary there is the need of a non-invasive device to measure respiratory volume to objectify complaints.

The ExSpiron© is a device for non-invasive monitoring of respiratory volume. The validation of this monitor in patients with ALS is the aim of this study.

The hypothesis is that the ExSpiron© delivers a valid assessment of respiratory volume in patients with ALS Objective: The primary objective is the validation of the ExSpiron© non-invasive monitor in patients diagnosed with ALS.

Study design: This is an intervention study The validation of the ExSpiron© in patients diagnosed with ALS is done during admission on the Respiratory Care Unit (RCU) of the University Medical Center Groningen (UMCG). At daytime, tidal volume (TV) and minute volume (MV) will be measured during spontaneous breathing with the ExSpiron© simultaneously with a pneumotachometer (gold-standard). After installation of the chest pad of the ExSpiron© and the pneumotachometer, the first measurements are in sitting position. Three complete cycles of ten breaths; normal breathing, slow-deep breathing and rapid-shallow breathing, will be done. Between each cycle, a pause is allowed. After completing this breathing sequence, it is repeated in supine position. If patients are not able to perform this in supine position, because of orthopnea, an angle of 45º degree is adequate. After completing this cycle, the chest pad should be left in place and the electromyography (EMG) equipment should be installed. During the first night of admission, a full night of measurement of TV and MV will be conducted using the ExSpiron©.

Study population: 10 patients diagnosed with ALS and an indication to start NIV, >18 years of age.

Intervention (if applicable): The ExSpiron© is a device for non-invasive monitoring of tidal volumes and minute ventilation in non-intubated patients by using a disposable chest pad.

Main study parameters/endpoints: The main endpoint is the validation of the ExSpiron© in patients diagnosed with ALS and screened positive for starting NIV.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: NIV has no known serious side effects. ALS patients differ in starting NIV is done on the RCU while patients are monitored as standard care, the ExSpiron© is not an extra risk complaints but those screened positive to start NIV are not associated with risks. The intervention product, ExSpiron© is a non-invasive monitor with a chest pad attached to the patient.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Participants diagnosed with ALS requiring NIV
* Age > 18 of age; < 85 years of age
* An indication to start chronic NIV, hypercapnic respiratory failure (arterial carbon dioxide PaCO2 > 6.0 kilo pascal (kPa) measured during daytime) or orthopnoea due to diaphragm paralysis.
* Participants are able to provide feedback
* Participants that are willing to participate and are able to consent and sign the informed consent form.

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in this study:
* Clinically unstable
* Acute respiratory failure
* Participants with refractory hypotension, defined as systolic blood pressure less than 90 mmHg, despite inotropic agents
* Uncontrolled cardiac ischemia or arrhythmias
* Participants suffering from metastatic or terminal cancer
* Other comorbid disease affecting respiration (ie obstructive sleep apnea, chronic obstructive pulmonary disease)
* Participants lacking functional medical decision-making

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The validity of the respiratory volumes (tidal volume and minute volume), compared tot the pneumotachometer. | 1 year
  The validation of the ExSpiron© non-invasive monitor in patients diagnosed with ALS.

SECONDARY OUTCOMES:
The BORG RPE score (Ratings of Percieved Exertion) | 1 year
  Visual analogue scale (VAS) score from 0-10, 0 is worse outcome, 10 is best outcome
The Amyotrophic lateral Sclerosis Assessment Questionnaire (ALSAQ-40) | 1 year
  questionaire, score 0-4; 0 is never and 4 is always or can not do.
SenTec is the name of a transcutaneous monitor | 1 year
  Gas exchange during the night with the transcutaneous monitor SenTec©
The EMG | 1 year
  Respiratory muscle activity and patient-ventilator asynchrony during the night and during NIV assessed with surface electromyograph

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wijkstra, prof, Principal Investigator — University Medical Center Groningen